CLINICAL TRIAL: NCT00212901
Title: Addition of Angiotensin Receptor Blockade to ACE Inhibition Versus High Dose ACE Inhibition for Reduction of Proteinuria in Patients With Diabetic Nephropathy
Brief Title: High Dose Ace Inhibitor Therapy Versus Combination of ACE and ARB Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2004482-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-07

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetes; Proteinuria; Angiotensin converting enzyme inhibitors; Angiotensin receptor antagonists
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Proteinuria

INTERVENTIONS:
Drug: High dose ACE-I vs ARB

SUMMARY:
Investigation of wheather addition of angiotensin receptor blocker (Irbesartan) to recommended doses of angiotensin converting enzyme inhibitor (trandolapril) is more effective in decreasing amount of protein in urine in patients with diabetic kidney disease than high doses of trandolapril.

ELIGIBILITY:
Inclusion Criteria:

1. Early diabetic nephropathy as defined by proteinuria between 500mg/24hr and 3g/24hr and GFR>50ml/min (as calculated by the Cockcroft-Gault formula), in the absence of clinical and laboratory evidence of other non-diabetic renal disease.
2. Controlled blood pressure (<150/<90)
3. Able to give informed consent
4. Between the ages of 18 and 75
5. Must be capable of providing a 24 hour urine collection
6. Negative BHcG test for ruling out pregnancy in women of childbearing age
7. Currently taking an angiotensin converting enzyme inhibitor

   -

Exclusion Criteria:

1. Creatinine clearance <50ml/min or 24hour protein excretion >3gm/d.
2. Hypotension as defined by the inability to add an ARB or increase ACE-I dose secondary to hypotensive symptomatology or a systolic Bp <100mmHg.
3. Serum potassium >5.5 on two separate occasions in the previous six months
4. Previous adverse reaction to angiotensin receptor antagonist medication
5. Use of NSAIDS including COX2 inhibitors
6. Pregnant or nursing women will be excluded
7. Currently taking an angiotensin receptor antagonist

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-08; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
reducing proteinuria

SECONDARY OUTCOMES:
glomerular filtration rate
side-effects of hypotension, postural symptom

CONTACTS AND LOCATIONS:
Overall Officials: Ayub Akbari, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada